CLINICAL TRIAL: NCT02026687
Title: Will Intrathecal Analgesia Contribute to a Faster Recovery Compared With Epidural Analgesia After Open Surgery for Gynecological Cancer. An Open Controlled Randomized Study.
Brief Title: Recovery and Analgesia After Surgery for Gynecological Cancer
Acronym: Speed
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lena Nilsson (Other)
Responsible Party: Sponsor-Investigator, Lena Nilsson, MD. PhD. Assoc professor., University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Speed
Record Dates: First submitted 2013-12-16; First posted 2014-01-03 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Gynecological Cancer
MeSH Terms: interventions — Injections, Epidural; Injections, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural analgesia (Active Comparator): The epidural anesthesia is applied at a low thoracic level, primarily Th10-Th11. A bolus dose of fentanyl together with a continuous infusion of bupivacain 2.5 mg/ml, fentanyl 1.8 µg/ml and epinephrine 2.5 µg/ml is used during surgery. Infusion rate is chosen by the attending anesthetist. Postoperatively the epidural anesthesia is continued until the morning of the third postoperative day using bupivacain 1 mg/ml, fentanyl 2 µg/ml and epinephrine 2µg/ml. Infusion rate is set by the responsible physician, maximum rate is 10 ml/hour.
  Interventions: Drug: Epidural
- Intrathecal analgesia (Experimental): The patient is given one intrathecal dose of plain bupivacaine (Marcain® spinal) 5 mg/ml, 15 mg together with morphine (Morphine Special®) 0,4 mg/ml, 0.2 mg and clonidine (Catapresan®) 150 µg/ml, 75 µg. The intrathecal mixture is given through a lumbal puncture at level L2/3, L3/4 or L4/5 before the induction of general anesthesia.
  Interventions: Drug: Intrathecal

INTERVENTIONS:
Drug: Epidural
  Arms: Epidural analgesia
Drug: Intrathecal
  Arms: Intrathecal analgesia

SUMMARY:
The purpose of the study is to compare epidural analgesia and intrathecal analgesia for explorative laparotomy through a middle-line incision for gynecological cancer in a fast track program to se if there is any difference in recovery. Length of stay is analyzed together with self-rate quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women with gynecological cancer (suspected or verified) planned for explorative laparotomy through a middle-line incision with a curative purpose.
* WHO performance status < 2.
* American Society of Anesthesiologists class 1-2.
* Women that understand and can express themselves in Swedish.
* Women that after verbal and written information accept participation in the study and have signed an informed consent.

Exclusion Criteria:

* Women where surgery is expected to include part/s, other than the abdominal surgery, where intrathecal or epidural analgesia is not expected to be effective
* Women with contra indications for intrathecal or epidural anesthesia.
* Women who are physically disabled and therefore nor expected to be mobilized on the day after surgery in the same way as non-disabled.
* Women with a mental retardation that makes it impossible to fill in the relevant questionnaires or makes it impossible to understand the meaning of participation, or if it is ethically doubtful to include the woman.
* Women with psychiatric or mental disorder that according to the responsible physician makes it unsuitable to participate in the study .

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Kjolhede P, Bergdahl O, Borendal Wodlin N, Nilsson L. Effect of intrathecal morphine and epidural analgesia on postoperative recovery after abdominal surgery for gynecologic malignancy: an open-label randomised trial. BMJ Open. 2019 Mar 4;9(3):e024484. doi: 10.1136/bmjopen-2018-024484. PMID 30837253

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Analgesia: The epidural anesthesia is applied at a low thoracic level, primarily Th10-Th11. A bolus dose of fentanyl together with a continuous infusion of bupivacain 2.5 mg/ml, fentanyl 1.8 µg/ml and epinephrine 2.5 µg/ml is used during surgery. Infusion rate is chosen by the attending anesthetist. Postoperatively the epidural anesthesia is continued until the morning of the third postoperative day using bupivacain 1 mg/ml, fentanyl 2 µg/ml and epinephrine 2µg/ml. Infusion rate is set by the responsible physician, maximum rate is 10 ml/hour.
  Epidural
- Intrathecal Analgesia: The patient is given one intrathecal dose of plain bupivacaine (Marcain® spinal) 5 mg/ml, 15 mg together with morphine (Morphine Special®) 0,4 mg/ml, 0.2 mg and clonidine (Catapresan®) 150 µg/ml, 75 µg. The intrathecal mixture is given through a lumbal puncture at level L2/3, L3/4 or L4/5 before the induction of general anesthesia.
  Intrathecal
Period: Overall Study
Arm/Group | Epidural Analgesia | Intrathecal Analgesia
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Analgesia | Intrathecal Analgesia | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (14.5) | 58.5 (8.5) | 58.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: From day of surgery (Day 0) until discharge after surgery
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 4 days
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Epidural: The EDA was performed by a low thoracic puncture. The epidural infusion included a bolus dose of fentanyl 50-100 µg and a bolus from a mixture of bupivacaine 2.4 mg/ml, adrenalin 2.4 µg/ml and fentanyl 1.8 µg/ml. For the EDA group, a continuous epidural infusion of a mixture of bupivacain 1 mg/ml + adrenalin 2µg/ml + fentanyl 2 µg/ml including the possibility of additional patient-controlled bolus doses was started postoperatively at the postoperative care unit and continued until the morning of the third postoperative day. The infusion rate, normally 4-8 ml/h, and bolus doses, normally 2 ml, were decided on by the responsible physician. The patients also had oral paracetamol 1330 mg three times daily, starting on the day of surgery. Oral oxycodone 10-20 mg twice daily and diclofenac 50 mg three times daily were added in the morning of the third postoperative day before removal of the epidural catheter according to the
- Spinal: The spinal group had an intrathecal combination of a single dose isobar bupivacaine 15 mg, morphine 0.2 mg and clonidine 75µg. The women in the ITM group received oral paracetamol 1330 mg and diclofenac 50 mg, both three times daily started on the day of surgery. Oxycodone 10-20 mg twice daily was added on the first postoperative day.
Arm/Group | Epidural | Spinal
Number analyzed (Participants) | 40 | 40
days | 4.3 [3.5 to 5.2] | 3.3 [3.1 to 4.8]

2. Secondary Outcome: Change in Quality of Life
Description: The questionnaire Short Form with 36 questions "SF-36" will be used preoperatively and at 6 weeks after surgery. The SF-36 consists of eight scaled subscores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental Health) and two Component summary scores (physical Component summary scoer, mental component summary score). A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Preoperatively and until 6 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Epidural | Spinal
Number analyzed (Participants) | 40 | 40
units on a scale
  SF-36 Physical component summary score baseline | 44 [34 to 53] | 45 [34 to 53]
  SF-36 Physical component summary score day 42 | 39 [34 to 44] | 38 [35 to 42]
  SF-36 mental component summary score baseline | 46 [35 to 52] | 46 [35 to 51]
  SF-36 mental component summary score day 42 | 49 [34 to 53] | 51 [39 to 55]

3. Other Pre Specified Outcome: Change in Pain
Description: Pain at rest will be assessed using a numeric rating scale from 0 (no pain) to 10 (worst imaginable pain). Pain is documented on the day of surgery (day 0), 3 times daily postoperative day 1, 2, 3, 4, 5, 6, 7, 14, 21, 28, 35 and 42.
  Scale: NRS Minimum value:0 Maximum value: 10. Higher scores indicate worse outcome.
Time Frame: Day of surgery (day 0) until 6 weeks after surgery
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Epidural | Spinal
Number analyzed (Participants) | 40 | 40
units on a scale
  Pain at rest Day 0 | 1.5 [0.8 to 2.1] | 2.7 [2.0 to 3.4]
  Pain at rest Day 1 | 1.6 [1.0 to 2.3] | 3.2 [2.6 to 3.8]
  Pain at rest Day 2 | 1.5 [0.9 to 2.1] | 2.1 [1.5 to 2.7]
  Pain at rest Day 3 | 2.9 [2.2 to 3.6] | 1.4 [0.8 to 2.1]
  Pain at rest Day 4 | 1.4 [0.8 to 1.9] | 1.6 [1.1 to 2.2]
  Pain at rest Day 5 | 1.1 [0.7 to 1.6] | 1.2 [0.7 to 1.7]
  Pain at rest Day 6 | 1.0 [0.5 to 1.4] | 1.1 [0.7 to 1.5]
  Pain at rest Day 7 | 1.1 [0.5 to 1.6] | 1.0 [0.6 to 1.3]
  Pain at rest Day 14 | 0.8 [0.4 to 1.2] | 0.7 [0.2 to 1.2]
  Pain at rest Day 21 | 0.5 [0.1 to 0.8] | 0.3 [0.0 to 0.6]
  Pain at rest Day 28 | 0.2 [0.0 to 0.3] | 0.2 [0.0 to 0.4]
  Pain at rest Day 35 | 0.3 [0.1 to 0.5] | 0.3 [0.0 to 0.6]
  Pain at rest Day 42 | 0.5 [0.0 to 0.9] | 0.1 [0.0 to 0.2]

ADVERSE EVENTS:
Arm/Group | Epidural | Spinal
Serious Adverse Events (participants affected / at risk) | 2/40 | 7/40
Other Adverse Events (participants affected / at risk) | 17/40 | 14/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural (N=40) | Spinal (N=40)
Intensive care treatment (Surgical and medical procedures) | 1 (1) | 1 (1)
Surgical intervention (Surgical and medical procedures) | 1 (1) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural (N=40) | Spinal (N=40)
Deviation from normal postoperative cause (Surgical and medical procedures) | 13 (13) | 8 (8)
Pharmacological treatment (Surgical and medical procedures) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No